CLINICAL TRIAL: NCT03442101
Title: Trajectories of Treatment Response as Window Into the Heterogeneity of Psychosis: a Longitudinal Multimodal Imaging Study in Medication-naïve First Episode Psychosis Patients
Brief Title: Trajectories of Treatment Response as Window Into the Heterogeneity of Psychosis: a Longitudinal Multimodal Imaging Study
Status: Active, not recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Dr. Adrianne C Lahti, Professor of Psychiatry, University of Alabama at Birmingham
Other Study IDs: IRB-300000959; R01MH113800 (NIH)
Record Dates: First submitted 2018-02-09; First posted 2018-02-22 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Antipsychotic drug plasma levels
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment group: These participants are newly diagnosed with psychosis.
  Interventions: Drug: Patients with psychosis will be treated with known antipsychotic medication

INTERVENTIONS:
Drug: Patients with psychosis will be treated with known antipsychotic medication — Subjects with first episode psychosis will be treated with risperidone, the most frequently used antipsychotic drug (APD) for 32 weeks. The study will follow a rigorous longitudinal design to capture treatment response whereby those without an adequate response after 16 weeks of treatment will be switched to aripiprazole, another APD for 16 weeks. All patients will be scanned four times: at baseline and after 6, 16, and 32 weeks of treatment.
  Other Names: Brain imaging scans will be obtained 4 times during the study

SUMMARY:
Psychosis is a heterogeneous disorder and present treatment only works for a limited number of patients. In order to identify new therapeutic targets, this study will longitudinally characterize the underlying pathologies in those with poor treatment response using complimentary brain imaging modalities.

DETAILED DESCRIPTION:
Schizophrenia is a heterogeneous disorder that likely involves multiple underlying pathological mechanisms, which has plagued attempts to identify rational therapeutic targets. All available antipsychotic drugs (APD) are dopamine receptor antagonists, but clinical response is variable, with a third of patients being partial responders, and a third non-responders. Arguably, those who respond well to APD have primarily dopaminergic abnormalities but it is imperative to also characterize the specific underlying pathologies in those with poor response in order to unravel the heterogeneity of psychosis and effectively develop new treatments. The investigators propose to longitudinally follow treatment response to APD for eight months in medication-naïve first episode psychosis (FEP) subjects using complementary brain imaging techniques.

The investigators have already identified provisional markers for several different pathophysiological mechanisms underlying psychosis, including abnormalities in glutamate, brain connectivity, and neurodevelopment that they can track with brain imaging. In addition, the investigators propose to study the changes that occur in the brain in early compared to delayed treatment responders and changes that occur over time in response to treatment. By characterizing treatment trajectories and their relationship to baseline pathophysiologic alterations, the investigators will further complement their mechanistic understanding of the heterogeneity of psychosis.

The investigators propose to study 117 well-characterized FEP subjects who are medication naïve and treat them with the most frequently used APD for 32 weeks. The investigators will follow a rigorous longitudinal design to capture treatment response whereby those without an adequate response after 16 weeks of treatment will be switched to another APD for 16 weeks. All patients will be scanned four times: at baseline and after 6, 16, and 32 weeks of treatment. The investigators will use (1) proton MR Spectroscopy (MRS), (2) task and resting state functional MRI and (3) MRI and diffusion weighted imaging (DWI) to measure brain biochemistry, function and structure. Using several imaging modalities has the potential to interrogate different neurobiological aspects of treatment response and will offer greater opportunities for clustering the patterns and combinations of the underlying pathologies in those with poor response.

Deconstructing the heterogeneity of psychosis has broad implications for the identification of specific targets for drug development, and to lay the groundwork needed to conduct therapeutic trials on patients characterized by their specific underlying psychopathology.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of first episode psychosis
* Never been treated with an antipsychotic medication
* Between the age of 17 and 35

Exclusion Criteria:

* Inability to sign informed consent assessed by the Evaluation to sign - - Consent form
* Poorly controlled acute or chronic medical and neurological conditions
* History of head trauma with loss of consciousness for >2 minutes
* Clinically significant depression, hypomania, or mania
* Active substance abuse or dependence (except for nicotine)
* Suspected substance-induced psychosis
* Treatment with drugs known to affect brain glutamate levels
* Pregnant females

Ages: 17 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: First episode psychosis subjects
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Measures of brain structure | 32 weeks
  Measures of brain structure, as measured with diffusion tensor imaging (DTI) that are associated at baseline (when patients are unmedicated) with subsequent treatment response to antipsychotic medication.
Measures of brain function | 32 weeks
  Measures of brain function, as measured with functional MRI (fMRI) that are associated at baseline (when patients are unmedicated) with subsequent treatment response to antipsychotic medication.
Measures of brain biochemistry | 32 weeks
  Measures of brain biochemistry, as measured with MR Spectroscopy, that are associated at baseline (when patients are unmedicated) with subsequent treatment response to antipsychotic medication.

SECONDARY OUTCOMES:
Changes in measures of brain structure | 32 weeks
  Changes in measures of brain structure over time that are associated with treatment response to antipsychotic medication.
Changes in measures of brain function | 32 weeks
  Changes in measures of brain function over time that are associated with treatment response to antipsychotic medication.
Changes in measures of brain biochemistry | 32 weeks
  Changes in measures of brain biochemistry over time that are associated with treatment response to antipsychotic medication.

OTHER OUTCOMES:
Trajectory of treatment response | 32 weeks
  Identification of clusters of participants following similar trajectories of treatment response over time, through measures of brain structure.
Trajectory of treatment response | 32 weeks
  Identification of clusters of participants following similar trajectories of treatment response over time, through measures of brain function.
Trajectory of treatment response | 32 weeks
  Identification of clusters of participants following similar trajectories of treatment response over time, through measures of brain biochemistry.

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne Lahti, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Sparks Center, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Maximo JO, Briend F, Armstrong WP, Kraguljac NV, Lahti AC. Salience network glutamate and brain connectivity in medication-naive first episode patients - A multimodal magnetic resonance spectroscopy and resting state functional connectivity MRI study. Neuroimage Clin. 2021;32:102845. doi: 10.1016/j.nicl.2021.102845. Epub 2021 Sep 29. PMID 34662778
- [Derived] Maximo JO, Nelson EA, Armstrong WP, Kraguljac NV, Lahti AC. Duration of Untreated Psychosis Correlates With Brain Connectivity and Morphology in Medication-Naive Patients With First-Episode Psychosis. Biol Psychiatry Cogn Neurosci Neuroimaging. 2020 Feb;5(2):231-238. doi: 10.1016/j.bpsc.2019.10.014. Epub 2019 Nov 9. PMID 31902581